CLINICAL TRIAL: NCT03960255
Title: Prospective Exploration of the Effect of Adiposity and Associated Microbial Factors on the Healing and Progression of Diabetic Foot Ulcers in Tanzania
Brief Title: Effect of Adiposity and Associated Local Microbial Factors on Healing and Progression of Diabetic Foot Ulcers
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Muhimbili University of Health and Allied Sciences (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Principal Investigator, Fredirick Mashili, Principal investigator, Muhimbili University of Health and Allied Sciences
Other Study IDs: DA.282/298/01.C/
Record Dates: First submitted 2019-05-20; First posted 2019-05-23 (Actual); Last update posted 2022-12-29 (Actual); Status verified 2022-12

CONDITIONS: Diabetic Foot Ulcer
Keywords: Adiposity; Diabetic foot ulcer; Anti-microbial resistance
MeSH Terms: conditions — Diabetic Foot; Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood specimen for biochemical measurements and wound biopsies for culture and sensitivity testing
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Normal adiposity group: Body fat < 25% and <32% in men and women respectively, will be categorized as high adiposity. This is according to the The American Council on Exercise criteria.
  Interventions: Other: Normal standard care
- High adiposity group: Body fat ≥ 25% and ≥32% in men and women respectively, will be categorized as high adiposity. This is according to the The American Council on Exercise criteria.
  Interventions: Other: Normal standard care

INTERVENTIONS:
Other: Normal standard care — Both groups will receive standardized treatment and care for diabetic foot ulcers

SUMMARY:
Diabetic foot ulcers (DFUs) and their associated complications like amputations are increasingly becoming a problem in low and middle income (LMI) countries. Obesity (increased body fat/adiposity), which has been shown to complicate many diseases, is also increasing in LMI setting. It is however not certain whether increased adiposity, may make it difficult for DFUs to heal. Investigators aim to understand whether increased adiposity and accompanied local microbial factors have any negative impact on healing and progression of DFUs.

DETAILED DESCRIPTION:
A prospective cohort of 300 individuals with type 2 diabetes presenting with diabetic foot ulcers (DFUs) at an outpatient clinic will be recruited. At baseline, participants will be stratified into normal and high adiposity groups as measured by Bioelectrical Impedance Analysis (BIA). Both groups will receive DFU management according to locally appropriate standards of care and followed-up for 24 weeks or until complete wound healing, whichever occurs first. Local microbial characteristics, presence or absence of infection and other clinical parameters will also be assessed, and compared between the two groups. Enrolling 150 participants per group will have a minimum power of 80% to detect a 20% difference in cumulative incidence of complete ulcer healing (at the 5% level of statistical significance) between the normal and high adiposity groups.

ELIGIBILITY:
Inclusion Criteria:

* History of type 2 diabetes mellitus (T2DM)
* Presence of participant's signed informed consent
* Age 30 years and above at the time the participant is signing the consent
* Tanzanians of African origin (Black Tanzanians)
* Presence of diabetic foot ulcer (DFUs) (new or recurrent)

Exclusion Criteria:

* Known patients with congestive cardiac and/or renal failure.
* Any patients with absolute or relative contraindication for tissue biopsy (for incident cases)
* Patients with obvious signs of gangrene
* DFU patients with non-healing ulcer of more than 52 weeks duration.
* DFU patients with below normal body mass index BMI (BMI below 18).

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants (males and females) will be newly reporting and known type 2 diabetes mellitus (T2DM) patients with diabetic foot ulcer (DFU) of any class, stage and grade (based on the university of Texas ulcer staging system). Any prior treatment and important information related to the ulcers and patients will be recorded using a pre-tested questionnaire. DFU will be defined as a full-thickness wound, through the dermis, below the ankle in an individual with T2DM. Duration of ulcers will be measured and reported in weeks. To recruit appropriate participants, a careful examination will be done with qualified and trained personnel. Prior to commencement of the study appropriate manuals and standard operating procedures will be prepared and used throughout the study period.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2021-02-20 (Actual); Primary Completion 2023-04-15 (Estimated); Study Completion 2023-05-20 (Estimated)

PRIMARY OUTCOMES:
Proportion (%) of patients with complete wound healing at 24 weeks | 24 weeks
  Complete healing will be defined based on the criteria of the wound healing society, as 100% re-epithelialization of the wound surface (complete wound closure) with a complete absence of drainage.

SECONDARY OUTCOMES:
Proportion of patients with worsening or improving ulcer progression (worsening of improving based on University of Texas ulcer grading system) | 24 weeks
  Proportion (%) of patients with unfavorable progression (worsening) of an ulcer to a more advanced stage/grade or favorable progression (improving) of an ulcer to an earlier stage/grade, among those enrolled into the study within the study time frame. The grades will be evaluated using the University of Texas ulcer grading system.
Proportion of patients ending up in amputation | 24 weeks
  Proportion (%) of patients getting amputations of a toe or foot on the same side as an index ulcer, among those enrolled into the study within the study time frame.
Proportion of patients who Die | 24 weeks
  Proportion (%) of patients who die among those enrolled into the study within the study time frame

CONTACTS AND LOCATIONS:
Locations (4):
- Tanzania (4):
  - Mnazi Mmoja Hospital, Zanzibar, Unguja
  - Abbas Medical Center, Dar es Salaam
  - Muhimbili Academic Medical Center, Dar es Salaam
  - Temeke regional hospital, Dar es Salaam

REFERENCES:
- [Derived] Mashili F, Joachim A, Aboud S, Mchembe M, Chiwanga F, Addo J, Kendall L, Ako A, Abbas Z. Prospective exploration of the effect of adiposity and associated microbial factors on healing and progression of diabetic foot ulcers in Tanzania: study protocol of a longitudinal cohort study. BMJ Open. 2019 Dec 16;9(12):e031896. doi: 10.1136/bmjopen-2019-031896. PMID 31848165